CLINICAL TRIAL: NCT06581783
Title: Impact of Timing of Premedication on Mucosal Visibility During Endoscopy
Brief Title: Impact of Timing of Premedication on Mucosal Visibility During Endoscopy-A Randomized Controlled Trial
Acronym: ENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Doctor, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: POMVDE
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-08

CONDITIONS: Endoscopy, Digestive System
MeSH Terms: interventions — Simethicone; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control (No Intervention): Normal endoscopic patients with out medication is required to compare with active groups.
- simethicone plus NAC combination time interval greater than 30 minutes (Experimental): Premixed medication (150mg) simethicone and 600mg nac with 100ml of water has to be given >30minutes for 273 patients.
  Interventions: Drug: Simethicone plus NAC
- simethicone plus NAC 10 to 20 minutes (Experimental): Premixed medication (150mg) simethicone and 600mg nac with 100ml of water has to be given 10-20 minutes time interval for 273 patients.
  Interventions: Drug: Simethicone plus NAC
- simethicone plus NAC 20 to 30 minutes (Experimental): Premixed medication (150mg) simethicone and 600mg nac with 100ml of water has to be given 20-30minutes for 273 patients.
  Interventions: Drug: Simethicone plus NAC

INTERVENTIONS:
Drug: Simethicone plus NAC — Drug simethicone plus N acetylcysteine will be given before endoscopy with different time intervals
  Other Names: placebo (water)
  Arms: simethicone plus NAC 10 to 20 minutes; simethicone plus NAC 20 to 30 minutes; simethicone plus NAC combination time interval greater than 30 minutes

SUMMARY:
UGI endoscopy(esophagogastroduodenoscopy) is the main diagnostic modality for direct visualization ,real time assessment and interpretation of findings encountered. The evaluation of esophagogastroduodenoscopy (EGD) quality measures encompasses several categories, such as structure, procedure, result, and adverse events. The peri-EGD period procedures fall under the procedural area, which is primarily concerned with preventing and minimising missed diagnoses.

. More aid in the identification and characterisation of gastrointestinal mucosal lesions is provided by endoscopes equipped with improved imaging technologies, such as multiband or narrow-band imaging (NBI). Despite these advancements of technological aspects, the unclean mucosal surface of the stomach can make these high-end pieces of equipment virtually useless To visualize properly and diagnose accurately there should be clear visibility of mucus apart from operator experience. Since the stage at diagnosis of upper gastrointestinal cancer is a major factor in survival, early detection is essential in improving the prognosis of patients the main factors responsible for hinderance of mucosal visibility are mucus foam and bubbles, which requires additional care for the clearance to enhance the vision and also decrease endoscopy duration by alleviating the need of repeated flushing and suctioning during endoscopy. The froth and bubbles are made of mucous secretions mixed with gastric juice and bile. Simethicone (polydimethylsiloxane and silicon dioxide) has been proven to be a promising defoaming agent as an endoscopic premedication in removing bubbles . Simethicone works by reducing the surface tension of air bubbles, and releases the trapped air by causing small bubbles to coalesce and collapse . N-acetylcysteine (nac), a mucolytic agent, has also been used as premedication acts by removing the mucous overlying the gastrointestinal mucosa 4-point scale described by Basford et al

1. No adherent mucus and clear views of the mucosa.
2. A thin coating of mucus that did not obscure views of the mucosa.
3. Some mucus/bubbles partially obscuring views of the mucosa (i. E. A small mucosal lesion might be missed without flushing
4. Heavy mucus/bubbles obscuring views of the mucosa (i. E. Extensive flushing is needed to avoid missing small mucosal lesions)

DETAILED DESCRIPTION:
Procedure

• Premixed medication (150mg simethicone and 600mg nac with 100ml of water) was given at specified timing Primary objective - comparison of mucosal visibility between 4 groups Secondary objectives - adverse events adequate gastric mucosal visibility lesion detection rate

ELIGIBILITY:
Inclusion Criteria:

Age >18years

Exclusion Criteria:

* History of upper gastrointestinal surgery
* Neurological disorders with impaired swallowing
* Active gastrointestinal bleeding,
* Caustic ingestion
* Pregnancy.
* Known history of multiple allergies
* Gastric outlet obstruction
* Esophageal motility disorders
* Contraindication for upper GI endoscopy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
comparison of mucosal visibility between 4 groups | 10-30 minutes
  Scores will be given based on Basford scale for esophagus, stomach (four parts: Cardia, fundus, body, antrum), Duodenum (D1, D2), score 1 indicates No adherent mucus and clear views of the mucosa, score 2 indicates A thin coating of mucus that did not obscure views of the mucosa, score 3 indicates some mucus/bubbles partially obscuring views of the mucosa score 4 indicates Heavy mucus obscuring views of the mucosa .

SECONDARY OUTCOMES:
To check adverse events during medication | 30 minutes
  adverse events may happen due to simethicone medicine like itching etc
To identify the lesion detection rate | 30 minutes
  During endoscopy procedure with different time intervals the lesions were noted

CONTACTS AND LOCATIONS:
Overall Officials: zaheer Dr Nabi, MBBS MD DNB, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology /Aig Hospitals, Hyderabad, Telangana, India